CLINICAL TRIAL: NCT06075628
Title: Long-Term Outcomes of Left Atrial Appendage Contrast Flow in CT Scans After Endocardial LAA Closure: The CF-CT Registry
Brief Title: Long-Term Outcomes of LAA Contrast Flow in CT Scans After Endocardial LAA Closure: The CF-CT Registry
Status: Recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRRF_CF-CT Registry_0021
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation; Ischemic Stroke, Acute
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amplatzer Amulet: This is the group of subjects who are implanted with Amplatzer Amulet device.
  Interventions: Other: Left Atrial Appendage Occlusion
- Watchman / Watchman FLX: This is the group of subjects who are implanted with Watchman / Watchman FLX device.
  Interventions: Other: Left Atrial Appendage Occlusion

INTERVENTIONS:
Other: Left Atrial Appendage Occlusion — Acute ischemic stroke is a major cause of morbidity and mortality in non-valvular Atrial Fibrillation (AF). Oral Anticoagulation (OAC) with Warfarin and Direct oral anticoagulants (DOACs) has been the mainstay to prevent systemic thromboembolism (STE) in this patient population. It is estimated that around 50% of patients who have AF with indication for OAC end up being not on OAC due to bleeding complications leaving them at high risk for developing STE. Left atrial appendage occlusion (LAAO) offers an option in such population.

SUMMARY:
This study is intended to assess the incidence and correlation to the development of peri-device leaks (PDLs), device related thrombosis (DRTs) and cerebral vascular accident (CVA)/transient ischemic attacks (TIAs) in association with left atrial appendage contrast flow (LAA-CF). It will be a multi-center, retrospective study. Approximately 100 subject charts will be reviewed.

DETAILED DESCRIPTION:
Although the clinical significance of long-term left atrial appendage contrast flow (LAA-CF) in computerized tomography (CT) scan is unknown, study by Lim et al reported that 45 days are not enough for complete left atrial appendage (LAA) seal-off after left atrial appendage occlusion (LAAO) in humans and anatomic closure may not necessarily ensure treatment success. Long-term monitoring is warranted in high-risk patients with LAAO after switching from anticoagulation to antiplatelet therapy. They reported possible explanations for residual LAA-CF after LAAO to be related to peri-device gaps, incomplete endothelialization on the device surface, an off-axis device, fabric leak through the non-endothelialized portion of the device.

To this date no studies or registries exist on long term follow up and association of Left Atrial Appendage Contrast Flow (LAA-CF). In this study with two FDA approved devices (Watchman/Watchman FLX and Amplatzer Amulet), it is hypothesized that the LAA contrast-flow (CF) rate is related to lack of endothelization of the implanted devices and potentially associated with peri-device leaks (PDLs), device related thrombosis (DRT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age.
* Subjects underwent LAA closure with Watchman/Watchman FLX or Amplatzer Amulet at our institution from January 2019 till June 2022

Exclusion Criteria:

* No definite exclusion criteria are defined for the study as all patients with Watchman-FLX or Amplatzer Amulet will be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Charts of all subjects who underwent LAA closure either with Watchman/Watchman FLX or Amplatzer Amulet device from January 2019 till June 2022 will be reviewed.
  Chart review will be performed up to 1 year, after the patient is discharged from the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and correlation to the development of Peri-Device Leak (PDLs), Device-Related Thrombus (DRT) or cerebral vascular accident (CVA) in association with LAA-CF | 12 Months
  Incidence and correlation to the development of PDLs, DRTs or CVA in association with LAA-CF will be assessed. These will be noted as either Yes or No.

SECONDARY OUTCOMES:
Total time to complete endothelization or no LAA-CF | 12 Months
  Total time to complete endothelization or no LAA-CF will be assessed.
Association of device size with LAA-CF | 12 Months
  Association of device size with LAA-CF will be assessed.
Association of landing zone with LAA-CF | 12 Months
  Association of landing zone with LAA-CF will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

REFERENCES:
- [Background] Dar T, Yarlagadda B, Vacek J, Dawn B, Lakkireddy D. Management of Stroke risk in atrial fibrillation patients with bleeding on Oral Anticoagulation Therapy-Role of Left Atrial Appendage Closure, Octreotide and more. J Atr Fibrillation. 2017 Dec 31;10(4):1729. doi: 10.4022/jafib.1729. eCollection 2017 Dec. PMID 29487685
- [Background] Viles-Gonzalez JF, Kar S, Douglas P, Dukkipati S, Feldman T, Horton R, Holmes D, Reddy VY. The clinical impact of incomplete left atrial appendage closure with the Watchman Device in patients with atrial fibrillation: a PROTECT AF (Percutaneous Closure of the Left Atrial Appendage Versus Warfarin Therapy for Prevention of Stroke in Patients With Atrial Fibrillation) substudy. J Am Coll Cardiol. 2012 Mar 6;59(10):923-9. doi: 10.1016/j.jacc.2011.11.028. PMID 22381428
- [Background] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Background] Meier B, Blaauw Y, Khattab AA, Lewalter T, Sievert H, Tondo C, Glikson M; Document Reviewers. EHRA/EAPCI expert consensus statement on catheter-based left atrial appendage occlusion. Europace. 2014 Oct;16(10):1397-416. doi: 10.1093/europace/euu174. Epub 2014 Aug 29. No abstract available. PMID 25172844
- [Background] Lim YM, Kim JS, Kim TH, Uhm JS, Shim CY, Joung B, Hong GR, Lee MH, Jang YS, Pak HN. Delayed left atrial appendage contrast filling in computed tomograms after percutaneous left atrial appendage occlusion. J Cardiol. 2017 Dec;70(6):571-577. doi: 10.1016/j.jjcc.2017.04.007. Epub 2017 May 22. PMID 28546017
- [Background] Whitlock RP, Healey JS, Holmes DR. Left atrial appendage occlusion debate revisited. Circulation. 2015 Feb 24;131(8):756-61. doi: 10.1161/CIRCULATIONAHA.114.008840. No abstract available. PMID 25712058